CLINICAL TRIAL: NCT03029208
Title: A 52-week Open-label (Sponsor-blind), Randomized, Active-controlled, Parallel-group, Multi-center Study to Evaluate the Efficacy and Safety of Daprodustat Compared to Recombinant Human Erythropoietin in Subjects With Anemia Associated With Chronic Kidney Disease Who Are Initiating Dialysis
Brief Title: Anemia Studies in Chronic Kidney Disease (CKD): Erythropoiesis Via a Novel Prolyl Hydroxylase Inhibitor (PHI) Daprodustat-in Incident Dialysis (ASCEND-ID)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201410; 2016-000507-86 (EudraCT Number)
Record Dates: First submitted 2017-01-20; First posted 2017-01-24 (Estimated); Results first posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Anaemia
Keywords: Daprodustat, recombinant human erythropoietin, darbepoetin, anemia, chronic kidney disease, dialysis, ESRD
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — GSK1278863; Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Daprodustat treated anemic subjects (Experimental): Subjects will receive oral daprodustat once daily.
  Interventions: Drug: Daprodustat; Drug: Iron therapy
- Darbepoetin alfa treated anemic subjects (Active Comparator): Subjects will receive darbepoetin alfa subcutaneously or intravenously.
  Interventions: Drug: Darbepoetin alfa; Drug: Iron therapy

INTERVENTIONS:
Drug: Daprodustat — Daprodustat will be supplied as film coated tablets for oral administration containing 1, 2, 4, 6, 8, or 10 mg of daprodustat. Doses of 12, 16, and 24 mg of daprodustat will be provided using multiples of these tablet strengths.
  Arms: Daprodustat treated anemic subjects
Drug: Darbepoetin alfa — Darbepoetin alfa will be supplied as prefilled syringes (PFS) for SC/IV injection available in strengths: 20, 30, 40, 60, 80, 100 and 150 mcg.
  Arms: Darbepoetin alfa treated anemic subjects
Drug: Iron therapy — Iron therapy will be administered if ferritin is <=100 ng/mL and/or TSAT is <=20%.

SUMMARY:
The purpose of this multi-center study is to evaluate the efficacy and safety of daprodustat in subjects with anemia associated with CKD.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 99 years of age inclusive.
* Planning to start chronic dialysis within the next 6 weeks (from the date of the screening visit) OR have started and received dialysis (as specified below) for end-stage renal disease for a maximum of <=90 days immediately prior to randomization and is not expected to stop dialysis during the duration of the trial: HD >=2 times per week or PD >=4 times per week including incremental schedule; subjects on continuous ambulatory peritoneal dialysis (CAPD) and automated peritoneal dialysis (APD) are eligible.
* Hemoglobin concentration as measured by HemoCue (range inclusive): 8 to 10.5 g/dL (5-6.5 millimoles per liter [mmol/L]) at screening and 8-11.0 g/dL (5 to 6.8 mmol/L) at randomization.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Planned living-related or living-unrelated kidney transplant during the study.
* Ferritin: <=100 nanograms per milliliter (ng/mL) (<=100 micrograms per liter [mcg/L]) at screening or after IV iron supplementation.
* Transferrin saturation (TSAT): <=20% at screening or after IV iron supplementation.
* Vitamin B12 (cobalamin): Below the lower limit of the reference range at screening or after vitamin B12 supplementation.
* Folate: <2.0 ng/mL (<4.5 nanomoles per liter [nmol/L]) at screening.
* Aplasias: History of bone marrow aplasia or pure red cell aplasia (PRCA).
* Other causes of anemia: Untreated pernicious anemia, thalassemia major, sickle cell disease, or myelodysplastic syndrome.
* Gastrointestinal (GI) bleeding: Evidence of actively bleeding gastric, duodenal, or esophageal ulcer disease or clinically significant GI bleeding <=10 weeks prior to screening through to randomization (Day 1).
* Use of any Erythropoiesis-stimulating agent (ESA) treatment within 8 weeks prior to screening except for limited use as part of dialysis initiation. Note : Limited use is defined as no more than 6 weeks of short acting ESA (rhEPO or biosimilars; maximum of 20000 unit total) or long acting ESA (darbepoetin alfa [maximum of 100 mcg total] or methoxy polyethylene glycol-epoetin beta [maximum of 125 mcg total]) received before or after starting dialysis.
* Myocardial infarction or acute coronary syndrome: <=10 weeks prior to screening through to randomization (Day 1).
* Stroke or transient ischemic attack: <=10 weeks prior to screening through to randomization (Day 1).
* Chronic Class IV heart failure, as defined by the New York Heart Association (NYHA) functional classification system.
* Current uncontrolled hypertension as determined by the Investigator that would contraindicate the use of rhEPO.
* QT correction using Bazett's (QTcB) (Day 1): QTcB >500 milliseconds (msec), or QTcB >530 msec in subjects with bundle branch block. There is no QTc exclusion for subjects with a predominantly ventricular paced rhythm.
* Liver disease (any one of the following): 1. Alanine transaminase (ALT) >2 times upper limit of normal (ULN) (screening only). 2. Bilirubin >1.5 times ULN (screening only) (NOTE: Isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). 3. Current unstable liver or biliary disease per investigator assessment, generally defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis. NOTE: Stable chronic liver disease (including asymptomatic gallstones, chronic hepatitis B or C, or Gilbert's syndrome) are acceptable if subject otherwise meets entry criteria.
* History of malignancy within the 2 years prior to screening through to randomization (Day 1), or currently receiving treatment for cancer, or complex kidney cyst (i.e. Bosniak Category II F, III or IV) >3 centimeter (cm). The only exception is localized squamous cell or basal cell carcinoma of the skin that has been definitively treated >=10 weeks prior to screening.
* History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational product or to darbepoetin alfa.
* Use of strong Cytochrome P4502C8 (CYP2C8) inhibitors (example gemfibrozil) or strong CYP2C8 inducers (example rifampin/rifampicin).
* Use of other investigational agent or device prior to screening through to randomization (Day 1). At screening, this exclusion applies to use of the investigational agent within 30 days or within five half-lives (whichever is longer).
* Any prior treatment with daprodustat for treatment duration of >30 days.
* Females only: Subject is pregnant [as confirmed by a positive serum human chorionic gonadotropin (hCG) test for females of reproductive potential (FRP) only], subject is breastfeeding, or subject is of reproductive potential and does not agree to follow one of the contraceptive options in the List of Highly Effective Methods for Avoiding Pregnancy.
* Any other condition, clinical or laboratory abnormality, or examination finding that the investigator considers would put the subject at unacceptable risk, which may affect study compliance (example intolerance to rhEPO) or prevent understanding of the aims or investigational procedures or possible consequences of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (103):
- United States (34):
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Cerritos, California
  - GSK Investigational Site, Escondido, California
  - GSK Investigational Site, Glendale, California
  - GSK Investigational Site, La Palma, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Lynwood, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Whittier, California
  - GSK Investigational Site, Middlebury, Connecticut
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Crystal Lake, Illinois
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Merrillville, Indiana
  - GSK Investigational Site, Michigan City, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lufkin, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Hampton, Virginia
- Argentina (9):
  - GSK Investigational Site, Ciudad Evita, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Morón, Buenos Aires
  - GSK Investigational Site, Pergamino, Buenos Aires
  - GSK Investigational Site, Pilar, Buenos Aires
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Formosa
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (3):
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, St Albans, Victoria
- Canada (3):
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
- Germany (3):
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Kaiserslautern, Rhineland-Palatinate
  - GSK Investigational Site, Wiesbaden
- India (9):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Delhi
  - GSK Investigational Site, Gūrgaon
  - GSK Investigational Site, Kozhikode
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Secunderabad
  - GSK Investigational Site, Thiruvananthapuram
- Italy (4):
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Cagliari, Sardinia
- Malaysia (3):
  - GSK Investigational Site, George Town
  - GSK Investigational Site, Ipoh
  - GSK Investigational Site, Kuala Lumpur
- Mexico (7):
  - GSK Investigational Site, Torreón, Coahuila
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Ciudad de México, State of Mexico
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, Aguascalientes
  - GSK Investigational Site, Tlalnepantla
- Poland (7):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Koło
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Ostrołęka
  - GSK Investigational Site, Ostróda
  - GSK Investigational Site, Szczecin
- Russia (6):
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Mytishchi
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Volzhskiy
- GSK Investigational Site, Cape Town, South Africa
- South Korea (5):
  - GSK Investigational Site, Anyang-Si, Gyeonggi-do
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon
- Spain (5):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Puerto Real
  - GSK Investigational Site, Seville
- United Kingdom (4):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Doncaster
  - GSK Investigational Site, London
  - GSK Investigational Site, Middlesbrough

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Singh AK, Cizman B, Carroll K, McMurray JJV, Perkovic V, Jha V, Johansen KL, Lopes RD, Macdougall IC, Obrador GT, Waikar SS, Wanner C, Wheeler DC, Wiecek A, Stankus N, Strutz F, Blackorby A, Cobitz AR, Meadowcroft AM, Paul G, Ranganathan P, Sedani S, Solomon S. Efficacy and Safety of Daprodustat for Treatment of Anemia of Chronic Kidney Disease in Incident Dialysis Patients: A Randomized Clinical Trial. JAMA Intern Med. 2022 Jun 1;182(6):592-602. doi: 10.1001/jamainternmed.2022.0605. PMID 35377393

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted across 14 countries. Participants were randomized to receive either Daprodustat or Darbepoetin alfa.
Pre-assignment Details: A total of 312 participants were randomized in the study.
Groups:
- Daprodustat: Participants received daprodustat film-coated tablets with titrated dose levels ranging from 1, 2, 4, 6, 8, 10, 12, 16, and 24 milligrams (mg) orally once daily for up to 52 weeks. Study treatment was dose-titrated to achieve and maintain hemoglobin (Hgb) in the target range (10 to 11 grams per deciliter [g/dL]).
- Darbepoetin Alfa: Participants received darbepoetin alfa as prefilled syringes (PFS) for subcutaneous or intravenous (IV) injection with 4-weekly total dose levels ranging from 20, 30, 40, 60, 80, 120, 160, 200, 300 and 400 microgram (mcg) for 52 weeks. Study treatment was dose-titrated to achieve and maintain Hgb in the target range (10 to 11 g/dL).
Period: Overall Study
Arm/Group | Daprodustat | Darbepoetin Alfa
Started | 157 | 155
Completed | 155 | 151
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daprodustat | Darbepoetin Alfa | Total
Number analyzed (Participants) | 157 | 155 | 312
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.7 (14.31) | 55.8 (15.70) | 54.7 (15.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 57 | 118
  Male | 96 | 98 | 194
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian (AI) or Alaskan Native (AN) | 5 | 2 | 7
  Asian: Central/South Asian Heritage | 7 | 6 | 13
  Asian: East Asian Heritage | 8 | 16 | 24
  Asian: South East Asian Heritage | 11 | 9 | 20
  Black or African American | 16 | 13 | 29
  White: Arabic/North African Heritage | 1 | 0 | 1
  White: White/Caucasian/European Heritage | 109 | 107 | 216
  Mixed race: AI or AN and White | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Hemoglobin (Hgb) During Evaluation Period (Week 28 to Week 52)
Description: Blood samples were collected from participants for Hgb measurement. Hgb during the evaluation period was defined as the mean of all available post-randomization Hgb values (on and off-treatment) during the evaluation period (Week 28 to Week 52). For the primary analysis missing post-Baseline Hgb values were imputed using pre-specified multiple imputations. Change from Baseline was defined as the average of post-randomization values during the evaluation period minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date. An analysis of covariance (ANCOVA) model including randomization stratification factors Baseline Hgb and treatment was performed to obtain a point estimate and two-sided 95 percent (%) confidence interval (CI) for the treatment difference (daprodustat-darbepoetin alfa).
Time Frame: Baseline (Pre-dose on Day 1) and evaluation period (Week 28 to Week 52)
Population: Intent-to-Treat (ITT) Population comprised all randomized participants (who received a treatment randomization number).
Measure: Least Squares Mean (Standard Error); unit: Grams per deciliter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 157 | 155
Grams per deciliter | 1.02 (0.086) | 1.12 (0.085)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Non-Inferiority — Non-inferiority was to be established if the lower limit of the two-sided 95% CI for the treatment difference was greater than the pre-specified non-inferiority margin of -0.75 g/dL; Least square (LS) mean difference = -0.10, 95% CI 2-sided [-0.34 to 0.14] — An ANCOVA model including randomization stratification factors Baseline Hgb and treatment was performed to obtain a point estimate and two-sided 95% CI for the treatment difference (daprodustat-darbepoetin alfa)

2. Secondary Outcome: Average Monthly Intravenous Iron Dose (Milligrams) From Baseline to Week 52
Description: Total IV iron dose per participant was calculated from Day 1 to the earliest of (Week 52 visit date, first blood [red blood cells or whole blood] transfusion date and treatment stop date plus [+] 1 day) which corresponds to the time while the participant was on randomized treatment and before receiving a blood transfusion. Average monthly IV iron dose was calculated by Total IV iron dose divided by (/) (the number of days from Day 1 to the earliest of [Week 52 visit date, first blood transfusion date and treatment stop date +1] /30.4375 days). Data for participants until they underwent a red blood cells or whole blood transfusion was included in the analysis.
Time Frame: Baseline (Day 1) to Week 52
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Milligram
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 156 | 154
Milligram | 144.7 (10.90) | 125.3 (10.97)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8949, ANCOVA; LS mean difference = 19.4, 95% CI 2-sided [-11.0 to 49.9] — An ANCOVA model was used to compare the difference in this average monthly IV iron dose between arms, including factors for Baseline dose, treatment and the randomization stratification factors

3. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP), Mean Arterial Blood Pressure (MAP) at Week 52
Description: SBP, DBP and MAP were measured in a semi-supine or seated position in the dialysis chair after at least a 5-minutes of rest. MAP is an average BP in an individual's arteries during a single cardiac cycle. Change from Baseline was calculated as post-dose visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date. This analysis was carried out by using mixed model repeated measures (MMRM) model.
Time Frame: Baseline (Day 1) and Week 52
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimeter of mercury
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 153 | 149
Millimeter of mercury
  SBP | -3.57 (2.063) | -6.80 (2.931)
  DBP | 0.21 (1.216) | -4.01 (1.650)
  MAP | -0.95 (1.364) | -5.05 (1.894)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8168, Mixed model repeated measures (MMRM); LS mean difference = 3.23, 95% CI 2-sided [-3.82 to 10.27] — The difference in change from Baseline in SBP at Week 52 was analyzed with a MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9793, MMRM; LS mean difference = 4.21, 95% CI 2-sided [0.17 to 8.26] — The difference in change from Baseline in DBP at Week 52 was analyzed with a MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms
Statistical Analysis 3: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9597, MMRM; LS mean difference = 4.10, 95% CI 2-sided [-0.51 to 8.70] — The difference in change from Baseline in MAP at Week 52 was analyzed with a MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms

4. Secondary Outcome: Change From Baseline in SBP, DBP, MAP at End of Treatment
Description: SBP, DBP and MAP were measured in a semi-supine or seated position in the dialysis chair after at least a 5-minutes of rest. MAP is an average BP in an individual's arteries during a single cardiac cycle. End of treatment value for the blood pressure parameters were defined as the latest value on or before the last non-zero dose date plus (+) 1 day. Change from Baseline was calculated as post-dose visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date. This analysis was carried out by using ANCOVA model.
Time Frame: Baseline (Day 1) and end of treatment (last on-treatment value until Week 52)
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Millimeter of mercury
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 154 | 153
Millimeter of mercury
  SBP | -3.23 (1.659) | -3.14 (1.664)
  DBP | 0.60 (1.016) | -1.39 (1.020)
  MAP | -0.68 (1.092) | -1.97 (1.096)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.4840, ANCOVA; LS mean difference = -0.09, 95% CI 2-sided [-4.72 to 4.53] — The difference in change from Baseline in SBP at the derived end of treatment was analyzed with an ANCOVA model including terms for treatment, prognostic randomization stratification factors
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9156, ANCOVA; LS mean difference = 1.99, 95% CI 2-sided [-0.85 to 4.82] — The difference in change from Baseline in DBP at the derived end of treatment was analyzed with an ANCOVA model including terms for treatment, prognostic randomization stratification factors
Statistical Analysis 3: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.7966, ANCOVA; LS mean difference = 1.29, 95% CI 2-sided [-1.76 to 4.33] — The difference in change from Baseline in MAP at the derived end of treatment was analyzed with an ANCOVA model including terms for treatment, prognostic randomization stratification factors

5. Secondary Outcome: Blood Pressure (BP) Exacerbation Events Rate Per 100 Participant Years
Description: BP exacerbation event is defined (based on post-dialysis BP) as SBP >=25 millimeter of mercury (mmHg) increased from Baseline or SBP >=180 mmHg; or DBP >=15 mmHg increased from Baseline or DBP >=110 mmHg. The BP exacerbation events per 100 participant years was estimated using the Negative Binomial Model.
Time Frame: Up to Week 52
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Number (95% Confidence Interval); unit: Events per 100 participant year
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 155 | 154
Events per 100 participant year | 352.50 [268.89 to 462.09] | 350.00 [267.72 to 457.56]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.5174, Negative binomial model; Ratio of exacerbation rate = 1.01, 95% CI 2-sided [0.73 to 1.39] — Model estimated exacerbation rates, ratio of model estimated exacerbation rates and CIs were estimated using a negative binomial model for the treatment group comparison

6. Secondary Outcome: Number of Participants With at Least One Blood Pressure Exacerbation Event During Study
Description: BP exacerbation was defined (based on post-dialysis BP) as: SBP >=25 mmHg increased from Baseline or SBP >=180 mmHg; DBP >=15 mmHg increased from Baseline or DBP >=110 mmHg. Number of participants with at least one blood pressure exacerbation event is presented.
Time Frame: Up to Week 52
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 155 | 154
Participants | 91 | 100

7. Secondary Outcome: Change From Baseline in Post-randomization Hgb at Week 52
Description: Blood samples were collected from participants for Hgb measurements. Change from Baseline was calculated as post-dose visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Day 1) and Week 52
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Grams per deciliter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 139 | 141
Grams per deciliter | 1.17 (0.117) | 1.13 (0.115)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; LS mean difference = 0.04, 95% CI 2-sided [-0.29 to 0.36] — The difference in change from Baseline in post-randomization Hgb at Week 52 was analyzed with a MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms

8. Secondary Outcome: Number of Hgb Responders (Hgb in the Analysis Range of 10 to 11.5 Grams/Deciliter) During Evaluation Period (Week 28 to Week 52)
Description: Mean Hgb during the evaluation period was defined as the mean of all evaluable Hgb values during the evaluation period (Week 28 to Week 52) including any evaluable unscheduled Hgb values that were taken during this time period. Hgb responders were defined as number of participants with a mean Hgb during the evaluation period that falls within the Hgb analysis range of 10-11.5 g/dL.
Time Frame: Weeks 28 to 52
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 133 | 133
Participants | 86 | 87
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.5411, Cochran-Mantel-Haenszel; Difference in response rate = -0.8, 95% CI 2-sided [-12.2 to 10.7] — A Cochran-Mantel-Haenszel (CMH) test adjusted for treatment and randomization stratification factors were used to compare the number of responders between the treatment groups

9. Secondary Outcome: Percentage of Time for Which Hgb Was Within the Analysis Range (10 to 11.5 g/dL) During Evaluation Period (Week 28 to Week 52): Non-inferiority Analysis
Description: Percentage of days for which a participant's Hgb was within the analysis range of 10-11.5 g/dL (both inclusive) during the evaluation period (Week 28 to Week 52), including any unscheduled evaluable Hgb values that were taken during this time period was calculated. Percentage of time for which Hgb was within range for a participant was calculated by dividing 'the total number of days that Hgb was within range during Weeks 28 to 52' by 'the total number of days the participant remained on treatment during Weeks 28 to 52'.
Time Frame: Weeks 28 to 52
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Percentage of days
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 128 | 129
Percentage of days | 57.0 [0.0 to 100.0] | 54.7 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Non-Inferiority — Non-inferiority was to be established if the lower limit of the two-sided 95% confidence interval for the treatment difference was greater than non-inferiority margin of -15%; Median Difference (Final Values) = 2.05, 95% CI 2-sided [-4.45 to 11.27] — Hodges-Lehmann Estimate of Treatment Difference has been reported

10. Secondary Outcome: Percentage of Time for Which Hgb Was Within the Analysis Range (10 to 11.5 g/dL) During Evaluation Period (Week 28 to Week 52): Superiority Analysis
Description: as for outcome 9
Time Frame: Weeks 28 to 52
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Percentage of days
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 128 | 129
Percentage of days | 57.0 [0.0 to 100.0] | 54.7 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.1538, van Elteren test; Probability = 0.54, 95% CI 2-sided [0.46 to 0.61] — Mann-Whitney estimate (Probability) of the treatment effect has been presented

11. Secondary Outcome: Number of Participants Permanently Stopping Randomized Treatment Due to Meeting Rescue Criteria
Description: Number of participants permanently stopping randomized treatment due to meeting rescue criteria has been presented.
Time Frame: Up to Week 52
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 157 | 155
Participants | 5 | 5
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Other; p = 0.5348, Wald test; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.31 to 3.66] — Hazard ratio was estimated using a Cox proportional hazard regression model adjusted for treatment group, dialysis type and dialysis start manner

12. Secondary Outcome: Change From Baseline in Physical Component Score (PCS) Using Short Form (SF)-36 Health-related Quality of Life (HRQoL) Questionnaire at Weeks 8, 12, 28, 52
Description: The SF-36 acute version 2 is a 36-item generic quality of life instrument designed to measure a participant's level of performance in the following 8 health domains: physical functioning, role-physical (role limitations caused by physical problems), social functioning, bodily pain, mental health, role-emotional (role limitations caused by emotional problems), vitality and general health. Each domain is scored from 0 (poorer health) to 100 (better health). The PCS is an average score derived from 4 domains (physical functioning, role-physical, bodily pain and general health) representing overall physical health. PCS ranges from 0 to 100; higher scores represent better health. Change from Baseline was calculated as post-dose visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Day 1), Weeks 8, 12, 28 and 52
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed (represented by n=X in the category titles).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 88 | 88
Scores on a scale
  Week 8, n=88,86: number analyzed (Participants) | 88 | 86
  Week 8, n=88,86 | 0.79 (0.648) | 1.18 (0.658)
  Week 12, n=88,88 | 1.67 (0.627) | 0.54 (0.631)
  Week 28, n=80,74: number analyzed (Participants) | 80 | 74
  Week 28, n=80,74 | 0.94 (0.697) | 0.45 (0.725)
  Week 52, n=67,65: number analyzed (Participants) | 67 | 65
  Week 52, n=67,65 | 0.61 (0.755) | 1.93 (0.774)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6641, MMRM; LS mean difference = -0.39, 95% CI 2-sided [-2.22 to 1.44] — SF-36 HRQoL PCS domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 8
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.1030, MMRM; LS mean difference = 1.13, 95% CI 2-sided [-0.63 to 2.89] — SF-36 HRQoL PCS domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 12
Statistical Analysis 3: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.3157, MMRM; LS mean difference = 0.49, 95% CI 2-sided [-1.51 to 2.48] — SF-36 HRQoL PCS domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 28
Statistical Analysis 4: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8855, MMRM; LS mean difference = -1.31, 95% CI 2-sided [-3.46 to 0.84] — SF-36 HRQoL PCS domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 52

13. Secondary Outcome: Change From Baseline in Mental Component Score (MCS) Using SF-36 HRQoL Questionnaire at Weeks 8, 12, 28, 52
Description: The SF-36 acute version 2 is a 36-item generic quality of life instrument designed to measure a participant's level of performance in the following 8 health domains: physical functioning, role-physical (role limitations caused by physical problems), social functioning, bodily pain, mental health, role-emotional (role limitations caused by emotional problems), vitality and general health. Each domain is scored from 0 (poorer health) to 100 (better health). MCS is an average score derived from 4 domains (vitality, social functioning, role-emotional and mental health) representing overall mental health. MCS ranges from 0 to 100; higher scores represent better health. Change from Baseline was calculated as post-dose visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Day 1), Weeks 8, 12, 28 and 52
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 88 | 88
Scores on a scale
  Week 8, n=88,86: number analyzed (Participants) | 88 | 86
  Week 8, n=88,86 | 0.10 (0.822) | 0.76 (0.839)
  Week 12, n=88,88 | 0.08 (0.813) | 1.60 (0.824)
  Week 28, n=80,74: number analyzed (Participants) | 80 | 74
  Week 28, n=80,74 | -0.02 (0.905) | 0.30 (0.942)
  Week 52, n=67,65: number analyzed (Participants) | 67 | 65
  Week 52, n=67,65 | -0.95 (1.029) | -0.72 (1.051)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.7146, MMRM; LS mean difference = -0.67, 95% CI 2-sided [-2.99 to 1.66] — SF-36 HRQoL MCS domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 8
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9050, MMRM; LS mean difference = -1.53, 95% CI 2-sided [-3.82 to 0.76] — SF-36 HRQoL MCS domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 12
Statistical Analysis 3: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.5950, MMRM; LS mean difference = -0.32, 95% CI 2-sided [-2.91 to 2.28] — SF-36 HRQoL MCS domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 28
Statistical Analysis 4: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.5619, MMRM; LS mean difference = -0.23, 95% CI 2-sided [-3.17 to 2.70] — SF-36 HRQoL MCS domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 52

14. Secondary Outcome: Change From Baseline in SF-36 HRQoL Scores for Bodily Pain, General Health, Mental Health, Role-Emotional, Role-Physical, Social Functioning at Weeks 8, 12, 28, 52
Description: The SF-36 acute version 2 is a 36-item generic quality of life instrument designed to measure a participant's level of performance in the following 8 health domains: bodily pain, general health, mental health, role-emotional (role limitations caused by emotional problems), role-physical (role limitations caused by physical problems), social functioning, physical functioning and vitality. Each domain is scored from 0 (poorer health) to 100 (better health). Each domain score ranges from 0 to 100, higher score indicates a better health state and better functioning. Change from Baseline was calculated as post-dose visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Day 1), Weeks 8, 12, 28 and 52
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 88 | 88
Scores on a scale
  Bodily pain: Week 8, n=88,86: number analyzed (Participants) | 88 | 86
  Bodily pain: Week 8, n=88,86 | -0.41 (0.833) | -0.55 (0.843)
  Bodily pain: Week 12, n=88,88 | -0.13 (0.892) | -0.06 (0.895)
  Bodily pain: Week 28, n=80,74: number analyzed (Participants) | 80 | 74
  Bodily pain: Week 28, n=80,74 | 1.08 (0.941) | -1.26 (0.976)
  Bodily pain: Week 52, n=67,65: number analyzed (Participants) | 67 | 65
  Bodily pain: Week 52, n=67,65 | -2.00 (1.084) | 0.61 (1.109)
  General health: Week 8, n=88,86: number analyzed (Participants) | 88 | 86
  General health: Week 8, n=88,86 | 0.80 (0.662) | 0.75 (0.674)
  General health: Week 12, n=88,88 | 0.87 (0.651) | 0.59 (0.658)
  General health: Week 28, n=80,74: number analyzed (Participants) | 80 | 74
  General health: Week 28, n=80,74 | 0.63 (0.693) | 0.37 (0.720)
  General health: Week 52, n=67,65: number analyzed (Participants) | 67 | 65
  General health: Week 52, n=67,65 | 0.40 (0.823) | 0.58 (0.841)
  Mental health: Week 8, n=88,86: number analyzed (Participants) | 88 | 86
  Mental health: Week 8, n=88,86 | -0.90 (0.825) | 0.25 (0.841)
  Mental health: Week 12, n=88,88 | 0.01 (0.707) | 1.42 (0.712)
  Mental health: Week 28, n=80,74: number analyzed (Participants) | 80 | 74
  Mental health: Week 28, n=80,74 | -0.69 (0.866) | -0.21 (0.902)
  Mental health: Week 52, n=67,65: number analyzed (Participants) | 67 | 65
  Mental health: Week 52, n=67,65 | -0.53 (0.994) | -0.27 (1.013)
  Role-emotional: Week 8, n=88,86: number analyzed (Participants) | 88 | 86
  Role-emotional: Week 8, n=88,86 | 0.83 (0.880) | 0.50 (0.896)
  Role-emotional: Week 12, n=88,88 | 0.55 (0.934) | -0.07 (0.946)
  Role-emotional: Week 28, n=80,74: number analyzed (Participants) | 80 | 74
  Role-emotional: Week 28, n=80,74 | 0.91 (0.929) | 0.39 (0.964)
  Role-emotional: Week 52, n=67,65: number analyzed (Participants) | 67 | 65
  Role-emotional: Week 52, n=67,65 | -1.60 (1.193) | -0.11 (1.216)
  Role-physical: Week 8, n=88,86: number analyzed (Participants) | 88 | 86
  Role-physical: Week 8, n=88,86 | 1.34 (0.806) | 2.64 (0.818)
  Role-physical: Week 12, n=88,88 | 2.39 (0.712) | 1.69 (0.716)
  Role-physical: Week 28, n=80,74: number analyzed (Participants) | 80 | 74
  Role-physical: Week 28, n=80,74 | 0.62 (0.799) | 1.49 (0.829)
  Role-physical: Week 52, n=67,65: number analyzed (Participants) | 67 | 65
  Role-physical: Week 52, n=67,65 | 1.49 (0.895) | 2.22 (0.913)
  Social functioning: Week 8, n=88,86: number analyzed (Participants) | 88 | 86
  Social functioning: Week 8, n=88,86 | 0.52 (0.929) | 1.55 (0.947)
  Social functioning: Week 12, n=88,88 | 0.98 (0.774) | 2.15 (0.783)
  Social functioning: Week 28, n=80,74: number analyzed (Participants) | 80 | 74
  Social functioning: Week 28, n=80,74 | 1.03 (0.943) | 0.95 (0.980)
  Social functioning: Week 52, n=67,65: number analyzed (Participants) | 67 | 65
  Social functioning: Week 52, n=67,65 | 0.39 (1.085) | -0.33 (1.105)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.4523, MMRM; LS mean difference = 0.14, 95% CI 2-sided [-2.21 to 2.49] — SF-36 HRQoL bodily pain domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 8
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.5222, MMRM; LS mean difference = -0.07, 95% CI 2-sided [-2.57 to 2.43] — SF-36 HRQoL bodily pain domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 12
Statistical Analysis 3: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.0440, MMRM; LS mean difference = 2.33, 95% CI 2-sided [-0.35 to 5.02] — SF-36 HRQoL bodily pain domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 28
Statistical Analysis 4: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9523, MMRM; LS mean difference = -2.61, 95% CI 2-sided [-5.68 to 0.46] — SF-36 HRQoL bodily pain domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 52
Statistical Analysis 5: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.4811, MMRM; LS mean difference = 0.05, 95% CI 2-sided [-1.82 to 1.91] — SF-36 HRQoL general health domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 8
Statistical Analysis 6: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.3834, MMRM; LS mean difference = 0.28, 95% CI 2-sided [-1.56 to 2.11] — SF-36 HRQoL general health domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 12
Statistical Analysis 7: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.3983, MMRM; LS mean difference = 0.26, 95% CI 2-sided [-1.72 to 2.24] — SF-36 HRQoL general health domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 28
Statistical Analysis 8: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.5617, MMRM; LS mean difference = -0.18, 95% CI 2-sided [-2.51 to 2.15] — SF-36 HRQoL general health domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 52
Statistical Analysis 9: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8336, MMRM; LS mean difference = -1.15, 95% CI 2-sided [-3.48 to 1.18] — SF-36 HRQoL mental health domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 8
Statistical Analysis 10: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9188, MMRM; LS mean difference = -1.41, 95% CI 2-sided [-3.40 to 0.57] — SF-36 HRQoL mental health domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 12
Statistical Analysis 11: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6495, MMRM; LS mean difference = -0.48, 95% CI 2-sided [-2.96 to 1.99] — SF-36 HRQoL mental health domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 28
Statistical Analysis 12: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.5737, MMRM; LS mean difference = -0.27, 95% CI 2-sided [-3.09 to 2.56] — SF-36 HRQoL mental health domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 52
Statistical Analysis 13: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.3963, MMRM; LS mean difference = 0.33, 95% CI 2-sided [-2.15 to 2.82] — SF-36 HRQoL role-emotional domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 8
Statistical Analysis 14: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.3220, MMRM; LS mean difference = 0.62, 95% CI 2-sided [-2.01 to 3.25] — SF-36 HRQoL role-emotional domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 12
Statistical Analysis 15: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.3485, MMRM; LS mean difference = 0.53, 95% CI 2-sided [-2.13 to 3.18] — SF-36 HRQoL role-emotional domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 28
Statistical Analysis 16: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8064, MMRM; LS mean difference = -1.49, 95% CI 2-sided [-4.87 to 1.90] — SF-36 HRQoL role-emotional domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 52
Statistical Analysis 17: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8687, MMRM; LS mean difference = -1.29, 95% CI 2-sided [-3.57 to 0.98] — SF-36 HRQoL role-physical domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 8
Statistical Analysis 18: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.2435, MMRM; LS mean difference = 0.71, 95% CI 2-sided [-1.29 to 2.70] — SF-36 HRQoL role-physical domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 12
Statistical Analysis 19: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.7747, MMRM; LS mean difference = -0.87, 95% CI 2-sided [-3.15 to 1.41] — SF-36 HRQoL role-physical domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 28
Statistical Analysis 20: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.7141, MMRM; LS mean difference = -0.73, 95% CI 2-sided [-3.26 to 1.81] — SF-36 HRQoL role-physical domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 52
Statistical Analysis 21: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.7803, MMRM; LS mean difference = -1.03, 95% CI 2-sided [-3.65 to 1.59] — SF-36 HRQoL social functioning domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 8
Statistical Analysis 22: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8556, MMRM; LS mean difference = -1.18, 95% CI 2-sided [-3.35 to 1.00] — SF-36 HRQoL social functioning domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 12
Statistical Analysis 23: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.4763, MMRM; LS mean difference = 0.08, 95% CI 2-sided [-2.61 to 2.77] — SF-36 HRQoL social functioning domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 28
Statistical Analysis 24: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.3208, MMRM; LS mean difference = 0.73, 95% CI 2-sided [-2.35 to 3.80] — SF-36 HRQoL social functioning domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 52

15. Secondary Outcome: Change From Baseline in Vitality Scores Using SF-36 HRQoL Questionnaire at Weeks 28, 52
Description: The SF-36 acute version 2 is a 36-item generic quality of life instrument designed to measure a participant's level of performance in the following 8 health domains: physical functioning, role-physical (role limitations caused by physical problems), social functioning, bodily pain, mental health, role-emotional (role limitations caused by emotional problems), vitality and general health. Each domain is scored from 0 (poorer health) to 100 (better health). Vitality ranges from 0 to 100; higher scores represent better health. Change from Baseline was calculated as post-dose visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Day 1), Weeks 28 and 52
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 80 | 74
Scores on a scale
  Week 28, n=80,74 | -0.08 (0.866) | 0.95 (0.902)
  Week 52, n=67,65: number analyzed (Participants) | 67 | 65
  Week 52, n=67,65 | 0.16 (0.907) | 1.61 (0.925)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.7910, MMRM; LS mean difference = -1.02, 95% CI 2-sided [-3.50 to 1.46] — SF-36 HRQoL vitality domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 28
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8648, MMRM; LS mean difference = -1.45, 95% CI 2-sided [-4.03 to 1.14] — SF-36 HRQoL vitality domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 52

16. Secondary Outcome: Change From Baseline in Physical Functioning Domain Scores Using SF-36 HRQoL Questionnaire at Weeks 28, 52
Description: The SF-36 acute version 2 is a 36-item generic quality of life instrument designed to measure a participant's level of performance in the following 8 health domains: physical functioning, role-physical (role limitations caused by physical problems), social functioning, bodily pain, mental health, role-emotional (role limitations caused by emotional problems), vitality and general health. Each domain is scored from 0 (poorer health) to 100 (better health). Physical functioning ranges from 0 to 100; higher scores represent better health. Change from Baseline was calculated as post-dose visit value minus (-) Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Day 1), Weeks 28 and 52
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 80 | 74
Scores on a scale
  Week 28, n=80,74 | 0.55 (0.863) | 0.83 (0.898)
  Week 52, n=67,65: number analyzed (Participants) | 67 | 65
  Week 52, n=67,65 | 0.14 (0.947) | 1.58 (0.973)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.5879, MMRM; LS mean difference = -0.28, 95% CI 2-sided [-2.75 to 2.19] — SF-36 HRQoL physical functioning domain score was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 28
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8525, MMRM; LS mean difference = -1.43, 95% CI 2-sided [-4.12 to 1.26] — SF-36 HRQoL physical functioning domain scor was analyzed using an MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms at Week 52

17. Secondary Outcome: Change From Baseline in Health Utility EuroQol 5 Dimensions 5 Level (EQ-5D-5L) Questionnaire Score at Week 52
Description: EQ-5D-5L consists of 2 concepts-EQ-5D-5L descriptive system and EQ Visual Analogue Scale (EQ-VAS). EQ-5D-5L is self-assessment questionnaire, consisting of 5items covering 5 dimensions (mobility,self care, usual activities, pain/discomfort and anxiety/depression). Each dimension is measured by 5-point Likert scale(no problems, slight problems, moderate problems, severe problems and extreme problems). Responses for 5 dimensions together formed a 5-figure description of health state(e.g.11111 indicates no problems in all 5 dimensions). Each of these 5 figure health states were converted to a single index score by applying country-specific value set formula that attaches weights to dimensions and levels. Range for EQ-5D-5L index score is -0.594 (worst health) to 1 (full health), higher the score better the health status. Change from Baseline was calculated as post-dose visit value-Baseline value. Baseline was latest non-missing pre-dose assessment on or before randomization date.
Time Frame: Baseline (Day 1) and Week 52
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 24 | 25
Scores on a scale | 0.00 (0.041) | -0.03 (0.040)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.3154, MMRM; LS mean difference = 0.03, 95% CI 2-sided [-0.09 to 0.14] — MMRM model was fitted from Baseline up to Week 52 with factors for treatment, time, dialysis type, dialysis start manner, Baseline value and Baseline value by time and treatment by time interactions

18. Secondary Outcome: Change From Baseline in EQ Visual Analogue Scale (EQ-VAS) at Week 52
Description: The EQ-5D-5L consists of 2 concepts -EQ-5D-5L descriptive system and EQ-VAS. The EQ-5D-5L is a self-assessment questionnaire, consisting of five items covering five dimensions (mobility, self care, usual activities, pain/discomfort and anxiety/depression). Each dimension is measured by a five-point Likert scale (no problems, slight problems, moderate problems, severe problems, and extreme problems). The range for the EQ-5D-5L index score is 0 to 1 with '0' is worst health and '1' is full health. The EQ VAS records the respondent's self-rated health on a vertical VAS, ranging from 0 to 100, where 0 represents the worst health one can imagine and 100 represents the best health one can imagine. Change from Baseline was calculated as post-dose visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Day 1) and Week 52
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 24 | 25
Scores on a scale | 3.4 (3.27) | 6.8 (3.28)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.7651, MMRM; LS mean difference = -3.4, 95% CI 2-sided [-12.7 to 5.9] — [estimate comment as in outcome 17, analysis 1]

19. Secondary Outcome: Change From Baseline in Chronic Kidney Disease- Anemia Symptoms Questionnaire (CKD-AQ) at Week 52
Description: CKD-AQ is 21-item patient reported outcome measure assessing symptoms and symptom impact in participants with anemia associated with CKD. It had 3 domains: 1.Tired/Low Energy/Weak scale consisting of 10 items; 2.Chest Pain/Shortness of Breath scale consisting of 4 items; and 3.Cognitive scale consisting of 3 items. The 4 CKD-AQ single items are: (shortness of breath, no activity), (severity-short breath, resting), (difficulty standing for long time) and (difficulty sleeping). Single-item were recorded based on a 0-100 scoring with 0=worst possible and 100=best possible score. Three domains scores were calculated as average of items in each domain and ranged from 0-100 where 0=worst possible and 100=best possible score. Change from Baseline was calculated as post-dose visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Day 1) and Week 52
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 76 | 80
Scores on a scale
  Tired/Low energy/Weak domain | -2.36 (2.007) | 4.07 (1.990)
  Chest pain/Shortness of breath domain | -1.83 (1.593) | 2.28 (1.557)
  Cognitive domain | -4.17 (1.893) | 2.43 (1.852)
  Shortness of breath, no activity | -1.90 (1.861) | 1.14 (1.826)
  Severity-short breath, Resting | -4.16 (1.869) | 0.12 (1.836)
  Difficulty standing for long time | -2.00 (2.812) | 3.30 (2.754)
  Difficulty sleeping | -5.27 (2.667) | 1.26 (2.611)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9875, MMRM; LS mean difference = -6.43, 95% CI 2-sided [-12.05 to -0.82] — Tired/Low energy/Weak domain: MMRM model was fitted from Baseline up to Week 52 with factors for treatment, time, dialysis type, dialysis start manner, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9663, MMRM; LS mean difference = -4.11, 95% CI 2-sided [-8.52 to 0.30] — Chest pain/Shortness of breath domain: MMRM model was fitted from Baseline up to Week 52 with factors for treatment, time, dialysis type, dialysis start manner, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 3: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9930, MMRM; LS mean difference = -6.60, 95% CI 2-sided [-11.84 to -1.35] — Cognitive domain: MMRM model was fitted from Baseline up to Week 52 with factors for treatment, time, dialysis type, dialysis start manner, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 4: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8765, MMRM; LS mean difference = -3.03, 95% CI 2-sided [-8.19 to 2.12] — Shortness of breath, no activity: MMRM model was fitted from Baseline up to Week 52 with factors for treatment, time, dialysis type, dialysis start manner, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 5: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9464, MMRM; LS mean difference = -4.27, 95% CI 2-sided [-9.48 to 0.94] — Severity-short breath, Resting: MMRM model was fitted from Baseline up to Week 52 with factors for treatment, time, dialysis type, dialysis start manner, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 6: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9101, MMRM; LS mean difference = -5.31, 95% CI 2-sided [-13.09 to 2.47] — Difficulty standing for long time: MMRM model was fitted from Baseline up to Week 52 with factors for treatment, time, dialysis type, dialysis start manner, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 7: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9586, MMRM; LS mean difference = -6.52, 95% CI 2-sided [-13.90 to 0.86] — Difficulty sleeping: MMRM model was fitted from Baseline up to Week 52 with factors for treatment, time, dialysis type, dialysis start manner, Baseline value and Baseline value by time and treatment by time interactions

20. Secondary Outcome: Change From Baseline in Patient Global Impression of Severity (PGI-S)
Description: The PGI-S is a 1-item questionnaire designed to assess participant's impression of disease severity on a 5-point disease severity scale (0=absent, 1=mild, 2=moderate, 3=severe, or 4=very severe). A higher score indicated worse outcome. Change from Baseline was calculated as post-dose visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Day 1), Weeks 8, 12, 28 and 52
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 100 | 103
Scores on a scale
  Week 8, n=100,100: number analyzed (Participants) | 100 | 100
  Week 8, n=100,100 | 0.16 (0.091) | -0.11 (0.092)
  Week 12, n=100,103 | 0.02 (0.077) | -0.03 (0.077)
  Week 28, n=92,85: number analyzed (Participants) | 92 | 85
  Week 28, n=92,85 | 0.09 (0.086) | -0.07 (0.089)
  Week 52, n=75,77: number analyzed (Participants) | 75 | 77
  Week 52, n=75,77 | 0.22 (0.106) | 0.04 (0.105)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9810, MMRM; LS mean difference = 0.27, 95% CI 2-sided [0.02 to 0.53] — MMRM model was fitted from Baseline up to Week 8 with factors for treatment, time, dialysis type, dialysis start manner, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6743, MMRM; LS mean difference = 0.05, 95% CI 2-sided [-0.17 to 0.26] — MMRM model was fitted from Baseline up to Week 12 with factors for treatment, time, dialysis type, dialysis start manner, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 3: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8997, MMRM; LS mean difference = 0.16, 95% CI 2-sided [-0.09 to 0.40] — MMRM model was fitted from Baseline up to Week 28 with factors for treatment, time, dialysis type, dialysis start manner, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 4: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8835, MMRM; LS mean difference = 0.18, 95% CI 2-sided [-0.12 to 0.47] — [estimate comment as in outcome 17, analysis 1]

21. Secondary Outcome: Plasma Concentration of Daprodustat (GSK1278863) and Its Metabolites GSK2391220 (M2), GSK2506104 (M3), and GSK2531401 (M13)
Description: Pharmacokinetic samples were collected at pre-dose, 0.5, 1, 2 and 3 hours post-dose on Week 4 or 8 or 12 for pharmacokinetic (PK) analysis of daprodustat (GSK1278863) and its metabolites GSK2391220 (M2), GSK2506104 (M3), and GSK2531401 (M13). GSK2391220, GSK2506104 and GSK2531401 are the metabolites of Daprodustat (GSK1278863). Protocol allowed participants to provide pharmacokinetic samples on Week 4 or 8 or 12. Pharmacokinetic Population comprised of participants for whom a pharmacokinetic sample was obtained and analyzed.
Time Frame: Pre-dose, 0.5, 1, 2 and 3 hours post-dose; each pharmacokinetic sample was taken at Week 4 or 8 or 12
Population: Pharmacokinetic Population. Only those participants with data available at the indicated time points were analyzed (represented by n=X in the category titles). Blood samples were not collected for PK analysis of daprodustat 12, 16 and 24 mg arms.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Groups:
- Daprodustat 1 mg: Participants received film-coated tablets of daprodustat 1 mg orally once daily for 52 weeks.
- Daprodustat 2 mg: Participants received film-coated tablets of daprodustat 2 mg orally once daily for 52 weeks.
- Daprodustat 4 mg: Participants received film-coated tablets of daprodustat 4 mg orally once daily for 52 weeks.
- Daprodustat 6 mg: Participants received film-coated tablets of daprodustat 6 mg orally once daily for 52 weeks.
- Daprodustat 8 mg: Participants received film-coated tablets of daprodustat 8 mg orally once daily for 52 weeks.
- Daprodustat 10 mg: Participants received film-coated tablets of daprodustat 10 mg orally once daily for 52 weeks.
- Daprodustat 12 mg: Participants received film-coated tablets of daprodustat 12 mg orally once daily for 52 weeks.
- Daprodustat 16 mg: Participants received film-coated tablets of daprodustat 16 mg orally once daily for 52 weeks.
- Daprodustat 24 mg: Participants received film-coated tablets of daprodustat 24 mg orally once daily for 52 weeks.
Arm/Group | Daprodustat 1 mg | Daprodustat 2 mg | Daprodustat 4 mg | Daprodustat 6 mg | Daprodustat 8 mg | Daprodustat 10 mg | Daprodustat 12 mg | Daprodustat 16 mg | Daprodustat 24 mg
Number analyzed (Participants) | 19 | 26 | 20 | 18 | 1 | 1 | 0 | 0 | 0
Nanogram per milliliter
  Daprodustat: Pre-Dose, n=19,26,20,18,1,1,0,0,0 | 2.118 (5.0030) | 1.015 (3.1451) | 0.5787 (1.5718) | 2.867 (6.6142) | 0.1030 (NA) — Standard deviation could not be calculated for single participant. | 0.1090 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  Daprodustat: 0.5 hour, n=19,26,20,18,0,1,0,0,0: number analyzed (Participants) | 19 | 26 | 20 | 18 | 0 | 1 | 0 | 0 | 0
  Daprodustat: 0.5 hour, n=19,26,20,18,0,1,0,0,0 | 5.675 (8.4998) | 4.664 (8.7508) | 10.27 (20.425) | 12.58 (23.742) |  | 145.0 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  Daprodustat: 1 hour, n=19,26,20,18,1,1,0,0,0 | 12.34 (13.435) | 21.45 (42.160) | 36.78 (62.497) | 45.48 (48.765) | 0.9120 (NA) — Standard deviation could not be calculated for single participant. | 79.60 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  Daprodustat: 2 hours, n=19,26,20,18,1,1,0,0,0 | 12.74 (9.9019) | 20.36 (22.210) | 54.68 (80.284) | 55.62 (51.471) | 32.00 (NA) — Standard deviation could not be calculated for single participant. | 27.60 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  Daprodustat: 3 hours, n=19,26,19,18,1,1,0,0,0: number analyzed (Participants) | 19 | 26 | 19 | 18 | 1 | 1 | 0 | 0 | 0
  Daprodustat: 3 hours, n=19,26,19,18,1,1,0,0,0 | 7.719 (5.9144) | 15.58 (13.694) | 43.34 (66.295) | 56.49 (74.357) | 25.30 (NA) — Standard deviation could not be calculated for single participant. | 11.00 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2391220: Pre-Dose, n=19,26,20,18,1,1,0,0,0 | 0.7106 (0.64028) | 2.124 (2.8721) | 2.087 (2.1371) | 3.560 (4.2255) | 4.450 (NA) — Standard deviation could not be calculated for single participant. | 6.560 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2391220: 0.5 hour, n=19,25,20,18,1,1,0,0,0: number analyzed (Participants) | 19 | 25 | 20 | 18 | 1 | 1 | 0 | 0 | 0
  GSK2391220: 0.5 hour, n=19,25,20,18,1,1,0,0,0 | 0.7602 (0.67950) | 1.807 (2.2007) | 1.822 (2.1355) | 2.410 (2.8243) | 3.950 (NA) — Standard deviation could not be calculated for single participant. | 6.740 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2391220: 1 hour, n=18,26,20,18,1,1,0,0,0: number analyzed (Participants) | 18 | 26 | 20 | 18 | 1 | 1 | 0 | 0 | 0
  GSK2391220: 1 hour, n=18,26,20,18,1,1,0,0,0 | 1.123 (0.76920) | 1.752 (1.8589) | 1.965 (2.2830) | 3.140 (2.4856) | 3.900 (NA) — Standard deviation could not be calculated for single participant. | 10.00 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2391220: 2 hours, n=19,26,20,18,1,1,0,0,0 | 1.745 (1.3160) | 2.969 (2.4659) | 4.008 (4.4522) | 6.336 (4.3723) | 4.700 (NA) — Standard deviation could not be calculated for single participant. | 16.20 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2391220: 3 hours, n=19,26,19,18,1,1,0,0,0: number analyzed (Participants) | 19 | 26 | 19 | 18 | 1 | 1 | 0 | 0 | 0
  GSK2391220: 3 hours, n=19,26,19,18,1,1,0,0,0 | 1.911 (1.2274) | 3.535 (2.7203) | 5.553 (6.5157) | 9.372 (6.6452) | 6.090 (NA) — Standard deviation could not be calculated for single participant. | 16.60 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2506104: Pre-Dose, n=19,26,20,18,1,1,0,0,0 | 1.270 (0.96071) | 3.508 (4.2066) | 3.879 (3.4207) | 5.921 (5.8981) | 8.710 (NA) — Standard deviation could not be calculated for single participant. | 9.500 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2506104: 0.5 hour, n=19,26,20,18,1,1,0,0,0 | 1.197 (0.85104) | 2.788 (2.9893) | 3.315 (3.4249) | 4.015 (3.7385) | 7.740 (NA) — Standard deviation could not be calculated for single participant. | 8.110 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2506104: 1 hour, n=19,26,20,18,1,1,0,0,0 | 1.364 (0.96292) | 2.610 (2.4761) | 3.268 (3.4808) | 4.333 (3.0505) | 7.460 (NA) — Standard deviation could not be calculated for single participant. | 12.40 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2506104: 2 hours, n=19,26,20,18,1,1,0,0,0 | 1.966 (1.3440) | 3.583 (2.8427) | 4.989 (5.2109) | 7.130 (4.5105) | 8.930 (NA) — Standard deviation could not be calculated for single participant. | 19.60 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2506104: 3 hours, n=19,26,19,18,1,1,0,0,0: number analyzed (Participants) | 19 | 26 | 19 | 18 | 1 | 1 | 0 | 0 | 0
  GSK2506104: 3 hours, n=19,26,19,18,1,1,0,0,0 | 2.190 (1.3898) | 4.145 (3.1757) | 6.503 (7.5130) | 9.942 (7.0616) | 10.10 (NA) — Standard deviation could not be calculated for single participant. | 22.00 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2531401: Pre-Dose, n=19,26,20,18,1,1,0,0,0 | 1.642 (1.4836) | 2.729 (1.8934) | 3.750 (3.8006) | 5.111 (4.0632) | 5.660 (NA) — Standard deviation could not be calculated for single participant. | 7.760 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2531401: 0.5 hour, n=19,26,20,18,1,1,0,0,0 | 1.427 (1.2870) | 2.170 (1.6621) | 3.263 (3.8737) | 3.800 (2.8722) | 4.960 (NA) — Standard deviation could not be calculated for single participant. | 6.460 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2531401: 1 hour, n=19,26,20,18,1,1,0,0,0 | 1.399 (1.4595) | 1.979 (1.6316) | 3.146 (4.0334) | 3.776 (3.4411) | 4.810 (NA) — Standard deviation could not be calculated for single participant. | 6.630 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2531401: 2 hours, n=19,26,20,18,1,1,0,0,0 | 1.690 (1.6309) | 2.338 (2.1467) | 3.711 (5.0223) | 4.892 (4.7877) | 5.190 (NA) — Standard deviation could not be calculated for single participant. | 8.290 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2531401: 3 hours, n=19,26,19,18,1,1,0,0,0: number analyzed (Participants) | 19 | 26 | 19 | 18 | 1 | 1 | 0 | 0 | 0
  GSK2531401: 3 hours, n=19,26,19,18,1,1,0,0,0 | 1.847 (1.7376) | 2.734 (2.6846) | 4.715 (7.2788) | 6.631 (7.1049) | 5.760 (NA) — Standard deviation could not be calculated for single participant. | 10.20 (NA) — Standard deviation could not be calculated for single participant. |  |  |

22. Secondary Outcome: Observed Concentration at Dosing Interval (Ctau) of Daprodustat (GSK1278863) and Its Metabolites GSK2391220 (M2), GSK2506104 (M3), and GSK2531401 (M13)
Description: Pharmacokinetic samples were collected at pre-dose, 0.5, 1, 2 and 3 hours post-dose on Week 4 or 8 or 12 for pharmacokinetic analysis of daprodustat (GSK1278863) and its metabolites GSK2391220 (M2), GSK2506104 (M3), and GSK2531401 (M13). GSK2391220, GSK2506104 and GSK2531401 are the metabolites of Daprodustat (GSK1278863). Protocol allowed participants to provide pharmacokinetic samples on Week 4 or 8 or 12.
Time Frame: Pre-Dose, 0.5, 1, 2 and 3 hours post-dose; each pharmacokinetic sample was taken at Week 4 or 8 or 12
Population: Pharmacokinetic Population. Only those participants with data available at the indicated time points were analyzed. Blood samples were not collected for PK analysis of daprodustat 12, 16 and 24 mg arms.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Daprodustat 1 mg | Daprodustat 2 mg | Daprodustat 4 mg | Daprodustat 6 mg | Daprodustat 8 mg | Daprodustat 10 mg | Daprodustat 12 mg | Daprodustat 16 mg | Daprodustat 24 mg
Number analyzed (Participants) | 19 | 26 | 20 | 18 | 1 | 1 | 0 | 0 | 0
Nanogram per milliliter
  Daprodustat | 2.118 (5.0030) | 1.015 (3.1451) | 0.5787 (1.5718) | 2.867 (6.6142) | 0.1030 (NA) — Standard deviation could not be calculated for single participant. | 0.1090 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2391220 | 0.7106 (0.64028) | 2.124 (2.8721) | 2.087 (2.1371) | 3.560 (4.2255) | 4.450 (NA) — Standard deviation could not be calculated for single participant. | 6.560 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2506104 | 1.270 (0.96071) | 3.508 (4.2066) | 3.879 (3.4207) | 5.921 (5.8981) | 8.710 (NA) — Standard deviation could not be calculated for single participant. | 9.500 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2531401 | 1.642 (1.4836) | 2.729 (1.8934) | 3.750 (3.8006) | 5.111 (4.0632) | 5.660 (NA) — Standard deviation could not be calculated for single participant. | 7.760 (NA) — Standard deviation could not be calculated for single participant. |  |  |

23. Secondary Outcome: Maximum Observed Concentration (Cmax) of Daprodustat (GSK1278863) and Its Metabolites GSK2391220 (M2), GSK2506104 (M3), and GSK2531401 (M13)
Description: as for outcome 22
Time Frame: Pre-Dose, 0.5, 1, 2 and 3 hours post-dose; each pharmacokinetic sample was taken at Week 4 or 8 or 12
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter
Arm/Group | Daprodustat 1 mg | Daprodustat 2 mg | Daprodustat 4 mg | Daprodustat 6 mg | Daprodustat 8 mg | Daprodustat 10 mg | Daprodustat 12 mg | Daprodustat 16 mg | Daprodustat 24 mg
Number analyzed (Participants) | 19 | 26 | 20 | 18 | 1 | 1 | 0 | 0 | 0
Nanogram per milliliter
  Daprodustat | 21.74 (10.998) | 32.29 (40.166) | 76.92 (81.867) | 100.2 (74.086) | 32.00 (NA) — Standard deviation could not be calculated for single participant. | 145.0 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2391220 | 2.160 (1.2596) | 4.139 (3.3561) | 5.780 (6.2840) | 10.36 (6.3377) | 6.090 (NA) — Standard deviation could not be calculated for single participant. | 16.60 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2506104 | 2.477 (1.3625) | 5.212 (4.5562) | 7.075 (7.1313) | 11.60 (6.8731) | 10.10 (NA) — Standard deviation could not be calculated for single participant. | 22.00 (NA) — Standard deviation could not be calculated for single participant. |  |  |
  GSK2531401 | 2.283 (1.8210) | 3.565 (2.6091) | 5.328 (6.9034) | 7.836 (6.6199) | 5.760 (NA) — Standard deviation could not be calculated for single participant. | 10.20 (NA) — Standard deviation could not be calculated for single participant. |  |  |

ADVERSE EVENTS:
Time Frame: All-cause mortality, treatment emergent non-serious adverse events and serious adverse events were collected up to follow-up visit (Week 58)
Description: Safety Population comprised of all randomized participants who received at least one dose of randomized treatment.
Arm/Group | Daprodustat | Darbepoetin Alfa
All-Cause Mortality (participants affected / at risk) | 17/157 | 12/155
Serious Adverse Events (participants affected / at risk) | 52/157 | 51/155
Other Adverse Events (participants affected / at risk) | 76/157 | 74/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daprodustat (N=157) | Darbepoetin Alfa (N=155)
Pneumonia (Infections and infestations) | 4 (7) | 7 (7)
Peritonitis (Infections and infestations) | 1 (1) | 3 (5)
Septic shock (Infections and infestations) | 2 (2) | 2 (2)
Post procedural infection (Infections and infestations) | 3 (3) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 3 (3)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal infection (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Clostridial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Device related bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 1 (1) | 0 (0)
Leptospirosis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 5 (9) | 3 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 3 (3)
Cardiac failure (Cardiac disorders) | 1 (1) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 4 (5)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Inadequate haemodialysis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Open globe injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Peritoneal dialysate leakage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Unintentional medical device removal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (7) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3)
Volvulus (Gastrointestinal disorders) | 1 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloody peritoneal effluent (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic gastropathy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (2) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 2 (2)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Uraemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (2)
Hypertensive urgency (Vascular disorders) | 1 (1) | 1 (1)
Lymphocele (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Steal syndrome (Vascular disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Sudden death (General disorders) | 2 (2) | 0 (0)
Catheter site haemorrhage (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 4 (4) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 2 (2)
Azotaemia (Renal and urinary disorders) | 1 (1) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Retinopathy hypertensive (Eye disorders) | 1 (1) | 0 (0)
Hydrocholecystis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daprodustat (N=157) | Darbepoetin Alfa (N=155)
Hypertension (Vascular disorders) | 27 (51) | 24 (35)
Dialysis hypotension (Vascular disorders) | 21 (34) | 15 (22)
Hypotension (Vascular disorders) | 7 (8) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 14 (17) | 10 (10)
Vomiting (Gastrointestinal disorders) | 11 (16) | 5 (5)
Nausea (Gastrointestinal disorders) | 8 (13) | 6 (6)
Nasopharyngitis (Infections and infestations) | 7 (12) | 9 (9)
Upper respiratory tract infection (Infections and infestations) | 7 (9) | 11 (12)
Catheter site infection (Infections and infestations) | 5 (5) | 8 (11)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 (12) | 9 (12)
Headache (Nervous system disorders) | 12 (14) | 9 (10)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 4 (4) | 8 (13)
Fluid overload (Metabolism and nutrition disorders) | 9 (9) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT03029208/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT03029208/SAP_001.pdf